CLINICAL TRIAL: NCT05297084
Title: Effect of Non Surgical Periodontal Treatment on Clinical Parameters and Gingival Crevicular Fluid Il-17 and Il-18 Levels in Aggressive Periodontitis Patients
Brief Title: Non Surgical Periodontal Treatment Effect on Il-17 and Il-18 in Aggressive Periodontitis
Status: Completed | Type: Observational
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Sarah Elkot, Lecturer of Oral Medicine, Periodontology and Diagnosis, Faculty of Oral and Dental Medicine, Future University in Egypt, Cairo, Egypt., Future University in Egypt
Other Study IDs: FUE11
Record Dates: First submitted 2022-03-02; First posted 2022-03-25 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Aggressive Periodontitis
Keywords: gingival crevicular fluid
MeSH Terms: conditions — Aggressive Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Periopaper strips stored in Eppendorf tubes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Aggressive periodontitis: 25 young medically free patients with deep periodontal pockets >5mm
  Interventions: Procedure: non surgical periodontal therapy
- Periodontally healthy individuals: 25 young medically free individuals with no periodontal inflammation signs

INTERVENTIONS:
Procedure: non surgical periodontal therapy — Scaling and root planing
  Groups: Aggressive periodontitis

SUMMARY:
clinical parameters and IL-17 and Il-18 GCF levels were measured in 25 aggressive periodontitis patients compared to 25 periodontally healthy individuals.

It was observed that that Clinical parameters and Il-17 and Il-18 levels are higher before treatment but decreased after treatment which suggests role of these interleukins in pathogenesis of aggressive periodontitis .

DETAILED DESCRIPTION:
Aggressive periodontitis is a type of rapidly progressing periodontal diseases .The three classic primary characteristics of this disease are ; occurring in young healthy patients with rapid attachment loss and familial aggregation .Bacteria-host interactions, insufficiencies in host defenses and possibly a genetic predisposition represent the etiologic factors . Beside the young age of onset, important factors as involvement of host factors and non-plaque-related etiologic factors have also been proposed .

Aim of the study:

Objectives were to compare and correlate the clinical parameters and biochemical parameters (Il-17 and Il-18 levels in GCF) of aggressive periodontitis patients (At baseline and after three months of nonsurgical treatment) versus periodontally healthy subjects at baseline.

Subjects and methods:

Populations included in the study:

A total of fifty individuals were enrolled and categorized as; group A that included twenty five aggressive periodontitis patients and group B which included twenty five periodontally healthy controls.

Clinical parameters:

Plaque index (PI) ,gingival index (GI), Probing pocket depth (PPD) and clinical attachment level (CAL) were measured at baseline for both groups and after three months of non surgical periodontal treatment completion for group A.

GCF sampling:

In group A ,the site with deepest probing depth was selected for GCF sampling while for group B , any site was sampled using PerioPaper strips .

Phase I periodontal treatment After baseline GCF sample collection and clinical measurement recordings, group A patients received phase I periodontal treatment.

Analysis of Il-17 and Il-18 levels in GCF:

GCF samples were examined by enzyme-linked immunosorbent assay (ELISA).Procedures were performed according to the directions in the kits.

ELIGIBILITY:
Inclusion Criteria:

-Medically free subjects.

Exclusion Criteria:

* Subjects with periodontal surgeries in the last 6 months.
* Subjects with prior use of antibiotics in the last 6 months.
* Smokers.
* Pregnant females.
* Lactating females.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Both genders Age between 18 and 30 years old
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-03-27 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Periopaper strips Il-17 and Il-18 GCF measurements | Change from Baseline Il-17 and Il-18 at 3 months
  measurement of Il-17 and Il-18 in GCF from aggressive periodontitis patients using periopaper strips

CONTACTS AND LOCATIONS:
Overall Officials: Sarah M Elkot, Lecturer, Principal Investigator — Lecturer of Oral Medicine and Periodontology
Locations (1):
- Faculty of oral and dental medicine,FUE, Cairo,Egypt, Cairo, Egypt